CLINICAL TRIAL: NCT04809974
Title: Randomized, Placebo-controlled Parallel Group Clinical Trial of Nicotinamide Riboside to Evaluate NAD+ Levels in Individuals With Persistent Cognitive and Physical Symptoms After COVID-19 Illness ("Long-COVID")
Brief Title: Clinical Trial of Niagen to Examine Recovery in People With Persistent Cognitive and Physical Symptoms After COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Edmarie Guzman-Velez, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P000158
Record Dates: First submitted 2021-03-19; First posted 2021-03-22 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Covid19; Sequelae of; Infection; Cognitive Symptom
Keywords: Niagen; vitamin B3; Long-COVID; Long-haulers; Dietary supplement
MeSH Terms: conditions — COVID-19; Infections; Neurobehavioral Manifestations; Post-Acute COVID-19 Syndrome | interventions — nicotinamide-beta-riboside; Niacinamide

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, parallel group, placebo-controlled design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo: 40 participants will take placebo in the form of a capsule.
  Interventions: Drug: Niagen
- Niagen (Experimental): Supplement: 60 participants will take Niagen 2000mg in the form of capsules daily.
  Interventions: Drug: Niagen

INTERVENTIONS:
Drug: Niagen — The intervention consists of taking Niagen and completing all tasks divided into 6 visits.
  Other Names: Nicotinamide Riboside; TruNiagen; Vitamin B3

SUMMARY:
The study will assess whether Niagen, a safe dietary supplement, improves recovery of COVID-19 related symptoms in individuals who were infected at least 2 months prior to study entry ("Long-COVID" "Long-haulers"). 60% of participants will receive Niagen and 40% will receive PBO. Outcomes will consist of standardized cognitive, neuropsychiatric, physical, functional and biomarker assessments.

DETAILED DESCRIPTION:
This study will recruit people who were infected with COVID-19 at least 2 months ago and continue to experience symptoms related to infection. Initially thought to be an acute illness like the flu, resulting in death for some or full recovery in most, scientists and clinicians are now appreciating that substantial numbers of COVID-19 illness survivors experience persistent, significant and sometimes disabling symptoms. Variously called "Long-COVID," "COVID long-haulers," or "chronic COVID syndrome", some of the most prominent symptoms are neurologic and neuropsychiatric, including cognitive impairment ('brain fog'), headache, fatigue, muscle aches and weakness, shortness of breath, hair loss and pain, among others. In this research study the investigators want to learn about whether taking Niagen (also known as Nicotinamide riboside, or NR), a daily supplement containing a form of Vitamin B3, can improve recovery of cognitive function, mood, and physical health in individuals who were infected with COVID-19 and continue to experience "brain fog" and other neurological and physical symptoms. The investigators think that this supplement may help improve thinking skills and other symptoms, and improve quality of life, in individuals who had COVID-19.

Participants will complete the following at baseline and every 5 weeks: 1) a standard cognitive battery and subjective cognitive complaints scales; 2) mood measures; 3) assessments of physical functioning, as well as of other common COVID-19-related symptoms; 4) blood draw; and 5) 2 optional MRIs. Participants will also wear a Fitbit and complete questionnaires to assess sleep and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* History of SARS-CoV-2 PCR+ at least 2 months prior to study entry;
* SARS-CoV-2 negative (PCR) at study entry;
* Persistent cognitive difficulties (esp. "brain fog") that began around the time of the acute COVID-19;
* At least two neurological and/or physical symptoms that started with COVID-19 infection and are ongoing at study entry, including fatigue, weakness, headache, loss of smell, tingling/numbness, shortness of breath, loss of appetite, palpitations/tachycardia, hair loss, musculoskeletal and/or chest pain;
* Willing and able to consent, complete all assessment and study procedures;
* Not pregnant or lactating.

Exclusion Criteria:

* Any specific central nervous system disease history (e.g. major clinical stroke, brain tumor, normal pressure hydrocephalus, etc);
* Clinically significant unstable medical condition that could affect safety or compliance with the study;
* Was intubated due to COVID-19;
* Major active or chronic unstable psychiatric illness (e.g. depression, bipolar disorder, obsessive compulsive disorder, schizophrenia) within the previous year;
* History of alcohol or other substance abuse or dependence within the past two years;
* Any significant systemic illness or medical condition that could affect safety or compliance with study;
* Current use of medications with psychoactive properties that may be deleteriously affecting cognition;
* Any known hypersensitivity to nicotinamide riboside, or its principal metabolite, nicotinamide mononucleotide;
* Use of other investigational agents or interventions one month prior to entry and for the duration of the trial;
* If participating in the optional magnetic resonance imaging (MRI) sub-study: Any contraindication to undergo MRI;
* Pregnant women or women who are planning to become pregnant within 7 months from study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-08-28 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2024-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edmarie Guzman-Velez, PhD, Principal Investigator — Massachusetts General Hospital and Harvard Medical School
Locations (1):
- Clinical Translational Research Unit, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu CY, Reynolds WC, Abril I, McManus AJ, Brenner C, Gonzalez-Irizarry G, Gutierrez-Martinez L, Sun O, Rosand J, Tanzi RE, Arnold SE, Guzman-Velez E. Effects of nicotinamide riboside on NAD+ levels, cognition, and symptom recovery in long-COVID: a randomized controlled trial. EClinicalMedicine. 2025 Nov 12;89:103633. doi: 10.1016/j.eclinm.2025.103633. eCollection 2025 Nov. PMID 41357333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between August 2021 and September 2023. They were recruited using flyers posted at Massachusetts General Hospital (main and Charlestown campuses), Partners Rally for Research, community events, physician referrals, and outreach to local institutions. Eligibility was assessed via telephone interview and an in-person screening visit.
Pre-assignment Details: 72 participants provided informed consent and completed an in-person screening visit. Eleven participants were deemed ineligible based on screening assessments and did not proceed. The remaining 61 participants entered a two-week placebo lead-in phase, during which 3 participants withdrew from the study. A total of 58 participants completed the lead-in phase, attended the baseline visit, and were randomized to study intervention.
Groups:
- Lead-in Phase: Participants assigned to the Lead-in Phase received placebo capsules at the screening visit and were instructed to take four capsules in the morning and four capsules in the evening (8 capsules daily) for two weeks. All capsules were visually identical to the active study drug and administered using the same dosing instructions as the randomized phase.
- Placebo: Participants randomized to the placebo group received placebo capsules twice daily for 10 weeks following a two-week placebo lead-in period. After the initial 10 weeks, participants crossed over to receive NR (TruNiagen, Chromadex) 1000 mg twice daily for an additional 10 weeks. Dosing was double-blinded. Participants completed assessments of cognitive, neuropsychiatric, physical, functional, and biomarker outcomes, along with actigraphy monitoring.
- Niagen: Participants randomized to the Niagen group received NR (TruNiagen, Chromadex) 1000 mg twice daily for 20 weeks following a two-week placebo lead-in period. Dosing was double-blinded. Participants completed assessments of cognitive, neuropsychiatric, physical, functional, and biomarker outcomes, along with actigraphy monitoring.
Period: Lead-in Phase
Arm/Group | Lead-in Phase | Placebo | Niagen
Started | 72 | 0 | 0
Screening | 72 | 0 | 0
Completed | 58 | 0 | 0
Not Completed | 14 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — No longer eligible | 11 | 0 | 0
Period: Randomized Phase
Arm/Group | Lead-in Phase | Placebo | Niagen
Started | 0 | 21 | 37
Baseline | 0 | 21 | 37
Visit 1 | 0 | 21 | 29
Visit 2 | 0 | 18 | 25
Visit 3 | 0 | 18 | 20
Visit 4 | 0 | 18 | 18
Follow-up | 0 | 17 | 15
Completed | 0 | 17 | 15
Not Completed | 0 | 4 | 22
Not completed — Lost to Follow-up | 0 | 1 | 5
Not completed — Met an exclusion criteria during the study (e.g., re-infected with COVID-19, started new medication) | 0 | 2 | 8
Not completed — Adverse Event | 0 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Niagen | Total
Number analyzed (Participants) | 21 | 37 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.76 (12.72) | 47.05 (13.79) | 45.86 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 26 | 42
  Male | 5 | 11 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 20 | 33 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 18 | 34 | 52
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: Participants]
  United States | 21 | 37 | 58
Education [Number; unit: Participants]
  High School/GED | 1 | 0 | 1
  Some College | 1 | 4 | 5
  Associate or Technical Degree | 0 | 6 | 6
  College | 8 | 21 | 29
  Professional Studies | 11 | 6 | 17

OUTCOME MEASURES:

1. Primary Outcome: Effect of Niagen on NAD+ and Cognitive Functioning
Description: Cognitive outcomes were assessed using the Everyday Cognition (ECog) scale, Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), and the Trail Making Test B (TMT-B). The ECog total score ranges from 39 to 156, and individual domain scores range from 1 to 4. Higher scores indicate greater subjective cognitive decline since COVID-19 infection. Individual RBANS index scores range from 40 to 160, and the Sum of Index Scores (sum of five index scores) ranges from 200 to 800. Higher index scores reflect better cognitive performance. The TMT-B score is the completion time in seconds, with a maximum time of 5 minutes. A lower time is indicative of a better performance. Change scores reflect the difference from Baseline to Week 10, and from Week 10 to Week 20. Positive change scores on the ECog indicate worsening subjective cognitive decline. Positive change scores on the RBANS indicate improvement. Positive change scores in the TMT-B represent worsening performance.
Time Frame: Baseline, Week 10 and Week 20
Population: Only participants with complete outcome data at both timepoints relevant to a given change score were included in the analysis. Participants with missing data at either timepoint were excluded from the analysis for that specific outcome. As a result, the number of participants analyzed is lower than the total number randomized in each group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Niagen | Placebo
Number analyzed (Participants) | 29 | 21
units on a scale
  ECog Total (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  ECog Total (Baseline to Week 10) | -0.104 (0.370) | -0.214 (0.370)
  ECog Total (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  ECog Total (Week 10 to Week 20) | -0.014 (0.548) | -0.147 (0.236)
  ECog Memory (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  ECog Memory (Baseline to Week 10) | -0.222 (0.422) | -0.285 (0.564)
  ECog Memory (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  ECog Memory (Week 10 to Week 20) | 0.068 (0.515) | -0.139 (0.498)
  ECog Language (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  ECog Language (Baseline to Week 10) | -0.216 (0.415) | -0.289 (0.378)
  ECog Language (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  ECog Language (Week 10 to Week 20) | 0.068 (0.528) | -0.088 (0.321)
  ECog Visualspatial (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  ECog Visualspatial (Baseline to Week 10) | 0.103 (0.564) | -0.203 (0.460)
  ECog Visualspatial (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  ECog Visualspatial (Week 10 to Week 20) | -0.132 (0.878) | -0.028 (0.283)
  ECog Planning (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  ECog Planning (Baseline to Week 10) | -0.130 (0.643) | -0.211 (0.478)
  ECog Planning (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  ECog Planning (Week 10 to Week 20) | 0.081 (0.642) | -0.089 (0.293)
  ECog Organization (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  ECog Organization (Baseline to Week 10) | 0.060 (1.014) | -0.100 (0.517)
  ECog Organization (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  ECog Organization (Week 10 to Week 20) | -0.179 (1.072) | -0.278 (0.423)
  ECog Attention (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  ECog Attention (Baseline to Week 10) | -0.150 (0.633) | -0.139 (0.479)
  ECog Attention (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  ECog Attention (Week 10 to Week 20) | -0.028 (0.808) | -0.347 (0.486)
  RBANS Sum of Index Scores (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  RBANS Sum of Index Scores (Baseline to Week 10) | 10.600 (29.819) | 10.000 (23.314)
  RBANS Sum of Index Scores (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  RBANS Sum of Index Scores (Week 10 to Week 20) | -8.111 (26.169) | -13.556 (40.441)
  RBANS Immediate Memory (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  RBANS Immediate Memory (Baseline to Week 10) | 5.800 (13.808) | 4.944 (12.085)
  RBANS Immediate Memory (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  RBANS Immediate Memory (Week 10 to Week 20) | -4.167 (11.784) | -6.389 (13.954)
  RBANS Delayed Memory (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  RBANS Delayed Memory (Baseline to Week 10) | 4.920 (11.420) | 2.167 (9.787)
  RBANS Delayed Memory (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  RBANS Delayed Memory (Week 10 to Week 20) | 0.944 (8.047) | -3.111 (12.925)
  RBANS Attention (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  RBANS Attention (Baseline to Week 10) | 4.080 (11.358) | 5.333 (12.825)
  RBANS Attention (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  RBANS Attention (Week 10 to Week 20) | -2.056 (12.822) | -0.389 (12.930)
  RBANS Language (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  RBANS Language (Baseline to Week 10) | -2.720 (12.674) | -0.222 (15.653)
  RBANS Language (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  RBANS Language (Week 10 to Week 20) | -1.833 (14.284) | -3.556 (16.639)
  RBANS Visuospatial (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  RBANS Visuospatial (Baseline to Week 10) | -1.560 (13.058) | -1.556 (12.538)
  RBANS Visuospatial (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  RBANS Visuospatial (Week 10 to Week 20) | 1.056 (14.198) | 0.167 (13.143)
  Trail-Making-Test B (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  Trail-Making-Test B (Baseline to Week 10) | -10.164 (21.456) | -6.574 (14.272)
  Trail-Making-Test B (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  Trail-Making-Test B (Week 10 to Week 20) | -3.525 (20.103) | -5.856 (19.148)

2. Secondary Outcome: Effect of Niagen on NAD+ and Depression Symptoms
Description: Depression symptoms were assessed using the Beck Depression Inventory (BDI), a 21-item self-report questionnaire measuring severity of depression symptoms. Total scores range from 0 to 63, with higher scores indicating more severe depression. Values represent mean change scores from Baseline to Week 10 and from Week 10 to Week 20.
Time Frame: Baseline, Week 10 and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Niagen | Placebo
Number analyzed (Participants) | 29 | 21
score on a scale
  BDI (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  BDI (Baseline to Week 10) | -1.360 (5.529) | 0.167 (5.659)
  BDI (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  BDI (Week 10 to Week 20) | 0.167 (4.301) | -2.111 (4.945)

3. Secondary Outcome: Effect of Niagen on NAD+ and Anxiety Symptoms
Description: Anxiety symptoms were assessed using the Beck Anxiety Inventory (BAI), a 21-item self-report questionnaire measuring severity of anxiety symptoms. Total scores range from 0 to 63, with higher scores indicating more severe anxiety. Values represent mean change scores from Baseline to Week 10 and from Week 10 to Week 20.
Time Frame: Baseline, Week 10 and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Niagen | Placebo
Number analyzed (Participants) | 29 | 21
score on a scale
  BAI (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  BAI (Baseline to Week 10) | -0.840 (7.301) | -1.333 (6.589)
  BAI (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  BAI (Week 10 to Week 20) | -0.167 (5.628) | -1.778 (4.387)

4. Secondary Outcome: Effect of Niagen on NAD+ and Other COVID-related Symptoms
Description: Fatigue was assessed using the Fatigue Severity Scale (FSS), a 9-item self-report measure with scores ranging from 1 to 7; higher scores indicate greater fatigue severity. Sleep quality was assessed using the Pittsburgh Sleep Quality Index (PSQI), a 19-item self-report measure with scores ranging from 0 to 21; higher scores indicate poorer sleep quality. All values represent mean change scores from Baseline to Week 10 and from Week 10 to Week 20.
Time Frame: Baseline, Week 10 and Week 20
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Niagen | Placebo
Number analyzed (Participants) | 29 | 21
score on a scale
  FSS Total Fatigue (Baseline to Week 10): number analyzed (Participants) | 25 | 18
  FSS Total Fatigue (Baseline to Week 10) | -3.400 (7.708) | -0.389 (8.417)
  FSS Total Fatigue (Week 10 to Week 20): number analyzed (Participants) | 18 | 18
  FSS Total Fatigue (Week 10 to Week 20) | 3.444 (9.083) | -4.278 (4.775)

ADVERSE EVENTS:
Time Frame: Adverse events were systematically collected at every visit, for a total of 24 weeks.
Groups:
- Lead in: Participants assigned to the Lead-in Phase received placebo capsules at the screening visit and were instructed to take four capsules in the morning and four capsules in the evening (8 capsules daily) for two weeks. All capsules were visually identical to the active study drug and were administered using the same dosing instructions as those in the randomized phase.
- Placebo: Participants randomized to the Placebo group took four capsules in the morning and four capsules in the evening (8 capsules daily) for 10 weeks following a two-week placebo lead-in period. After the initial 10 weeks, participants crossed over to receive 1000 mg of NR (Niagen) twice daily for an additional 10 weeks. Dosing was double-blinded. Participants completed clinical assessments and cognitive testing at baseline, Visit 2, and Visit 4, and provided blood at every visit since baseline.
- Niagen: Participants randomized to the NR group received 1000 mg of NR (Niagen) twice daily for 20 weeks following a two-week placebo lead-in period. Dosing was double-blinded. Participants completed clinical assessments and cognitive testing at baseline, Visit 2, and Visit 4, and provided blood at every visit since baseline.
Arm/Group | Lead in | Placebo | Niagen
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/21 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/21 | 1/37
Other Adverse Events (participants affected / at risk) | 1/72 | 19/21 | 25/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead in (N=72) | Placebo (N=21) | Niagen (N=37)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to Niagen: One serious adverse event (suicidal ideation) occurred in the Niagen group. This event was deemed unrelated to the study drug or procedures by the participant and several licensed clinicians.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lead in (N=72) | Placebo (N=21) | Niagen (N=37)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) — 1 possibly related in placebo group; 1 not related in Niagen group.
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) — 2 not related in Niagen group.
Arm pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Back spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — 1 not related in placebo group.
Brusing (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — 1 probably related in placebo group.
Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Cold hands (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — 1 not related in placebo group.
Cold Sweats (General disorders) | 0 (0) | 1 (1) | 0 (0) — 1 possibly related in placebo group.
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — 1 not related in placebo group.
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — 1 not related in Niagen group; 1 possibly related in placebo group.
COVID-19 infection (Infections and infestations) | 0 (0) | 1 (1) | 4 (4) — 4 not related in Niagen group; 1 not related in placebo group.
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) — 1 not related in Niagen group; 1 not related in placebo group
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) — 1 possibly related in placebo group; 1 possibly related in Niagen group.
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — 1 possibly related in Niagen group.
Edema of hand (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Edema of leg (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Facial flushing (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) — 1 possibly related and 1 probably related in Niagen group.
Facial pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) — 1 possibly related in placebo group and 1 not related in Niagen group.
Falx cerebri calcification (Investigations) | 0 (0) | 1 (1) | 0 (0) — 1 not related in placebo group.
GI discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (4) — 1 possibly related in placebo group; 1 possibly related and 3 not related in Niagen group.
Hand trembling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) — 1 probably related in Niagen group; 2 possibly related in placebo group
Heartburn (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) — 2 possibly related in placebo group.
Worsening IBS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — 1 possibly related in Niagen group.
Increased eructation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — 1 possibly related in placebo group.
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — 1 not related in placebo group.
Injury (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) — 3 not related in placebo group.
Joint ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — 1 possibly related in placebo group.
Kidney stone (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — 1 not related in placebo group.
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) — 1 probably related and 1 not related in Niagen group.
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — 1 definitely related in Niagen group.
Low vitamin B12 (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) — 1 possibly related in placebo group.
Muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — 1 probably related in placebo group.
Muscle strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) — 2 not related in placebo group.
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) — 1 definitely, 1 probably, and 1 possibly related in Niagen group; 1 probably and 1 possibly related in placebo group.
Night sweats (General disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Nocturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — 1 not related in placebo group.
Otitis media (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Paresthesia in extremities (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — 1 possibly related in Niagen group.
Paroxysmal blood pressure (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) — 1 not related in lead in group.
Pineal cyst (Investigations) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) — 2 not related in Niagen group.
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) — 1 definitely, 2 possibly, and 1 not related in Niagen group.
Sinus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) — 1 not related in Niagen group; 1 not related in placebo group.
Restless leg (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Stiffness in finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) — 1 possibly related in Niagen group.
Upper respiratory infection (Infections and infestations) | 0 (0) | 4 (4) | 6 (7) — 7 not related in Niagen group; 4 not related in placebo group.
Urine odor (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Vertigo (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) — 1 definitely and 1 not related in Niagen group; 1 not related in placebo group.
Viral syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — 1 not related in Niagen group.
Worsening bile reflux (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — 1 possibly related in placebo group.
Worsening cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — 1 not related in placebo group.
Worsening insomina (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) — 2 not related in Niagen group.
Worsening sleep (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (2) — 1 possibly related and 1 not related in Niagen group; 1 not related in placebo group.

LIMITATIONS AND CAVEATS:
The sample size of individuals who completed the clinical trial was relatively small, and COVID-19 infection status was based on self-report. Moreover, we exclusively included individuals experiencing brain fog, preventing us from assessing whether NR could be beneficial for those with different long-COVID symptom profiles.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT04809974/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/74/NCT04809974/ICF_001.pdf